CLINICAL TRIAL: NCT06808581
Title: EVALUATION OF SERUM INFLAMMATORY CYTOKINE CONCENTRATION
Brief Title: EVALUATION OF SERUM INFLAMMATORY CYTOKINE CONCENTRATION IN HEREDITARY SENSITIVOMOTOR NEUROPATHIES
Acronym: CytokinesUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-AOI-04
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Charcot-Marie-Tooth Disease; Hereditary Neuropathy With Hypersensitivity to Pressure
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identify a circulating marker of inflammation in patients with CMT or HNPP (Experimental): CMT = Charcot-Marie-Tooth disease HNPP = hereditary neuropathy with hypersensitivity to pressure
  Interventions: Diagnostic Test: blood test for pro-inflammatory cytokines and ultrasound of the median nerves

INTERVENTIONS:
Diagnostic Test: blood test for pro-inflammatory cytokines and ultrasound of the median nerves — Blood test and ultrasound

SUMMARY:
The most common forms of hereditary neuropathy are Charcot-Marie-Tooth disease (CMT) and hereditary neuropathy with hypersensitivity to pressure (HNPP) or tomacular neuropathy. A number of patients with one of these pathologies have inflammatory infiltrates in their nerves. Although the pathophysiology has not yet been well understood, the involvement of the immune system has been discussed. Nerve hypertrophy is the main anomaly described in ultrasound in demyelinating hereditary neuropathies and to a lesser extent in axonal forms. Investigators propose to understand if there is a circulating marker of inflammation in patients with CMT or HNPP and find a correlation between the increase in plasma pro-inflammatory cytokines and ultrasound changes.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patient over 18 years of age
* Patient with CMT of HNPP with genetic confirmation, or acquired acute inflammatory disease such as Guillain-Barré syndrome
* Patient able to walk alone or with a walking aid.
* Patient affiliated to a social security scheme,
* Patient who has given his consent in writing after written and oral information

Inclusion Criteria for Healthy Volunteers:

* Patient over 18 years of age
* Patient affiliated to a social security scheme,
* Patient who has given his consent in writing after written and oral information -

Exclusion Criteria:

* Subject protected by law under guardianship or curators, or not able to participate in a clinical study under article L. 1121-16 of the French Public Health Code;
* Subject who has participated in a clinical research study during the last 3 months where he/she was exposed to a pharmaceutical product or medical device;
* Subject who has stayed in a tropical or subtropical country during the last 3 months;
* Pregnant or breastfeeding subject for women of childbearing age;
* Subject who has been physically active for less than 10 hours;
* Subject on a particular diet for medical reasons and prescribed by a doctor or dietitian (e.g., low-calorie or cholesterol-lowering diet);
* Person who regularly consumes large amounts of alcohol, i.e. more than 50 g of pure alcohol per day (for example, more than 4 glasses of wine 150 ml, more than 4 beers 250 ml, or more than 4 glasses of 40 ml containing a strong alcohol);
* Person who has used an illicit recreational drug in the last 3 months;
* Subject who has taken an immunosuppressive or immunomodulatory drug (except for intranasal or topical corticosteroids) in the last 2 weeks, or for more than 14 consecutive days in the last 6 months;
* Subject who has been vaccinated in the last 3 months;
* Subject who received a blood transfusion or immunoglobulins in the last 3 months;
* Person reporting not having fasted for at least 10 hours;
* Person reporting human immunodeficiency virus, hepatitis B virus or hepatitis C virus ;
* Subject who has had an infectious episode in the 3 weeks preceding the visit;
* Test positive for pregnancy urine;
* Subject with severe and/or chronic and/or recurrent disease
* Subject diagnosed with cancer and not in remission for more than 5 years.
* (only for patients) Other associated peripheral nerve pathology already diagnosed (inherited neuropathy or acquired neuropathy from another etiology).
* (only for Health volunteers) Presence of functional or physical signs of involvement of the median nerves, ulnar, external Sciatica Poplitea, internal Sciatica Poplitea, sural

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Compare serum interleukin IL-1β between different subgroups of patients with genetic neuropathy (demyelinating/axonal/intermediate Charcot-Marie-Tooth disease (CMT) and hereditary neuropathy with hypersensitivity to pressure (HNPP)) and a control group. | at inclusion
  Serum interleukin IL-1β will be measured using v-plex MSD (Meso Scale Discovery) technology. The IL-1β concentrations will be expressed in ng/ml by calibration with a standard range

SECONDARY OUTCOMES:
Compare the serum concentration of pro-inflammatory cytokines among the different subgroups of patients with genetic neuropathy (demyelinating/axonal/intermediate CMT, HNPP) and with a homogeneous group of control subjects. | at inclusion
  A blood sample for measuring inflammatory cytokines (interleukins IL-6, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-7, IL-8, IL-10, IL-12 p70, IL-12/IL-23 p40, IL-13, IL-15, IL-16, IL-17A, interferon γ, Tumor necrosis factor α and β, Granulocyte-Macrophage Colony-Stimulating Factor, vascular endothelial growth factor, Chemokines CCL2, CCL3, CCL4, CCL11, CCL13, CCL17, CCL22, CCL26, and CXCL10) using v-plex technology (MesoScale Discovery)
Compare morphological characteristics obtained by high-frequency ultrasound between the different subgroups of subjects | within 2 months after inclusion
  The descriptive analysis of the morphology of the nerves will be carried out using a high-frequency ultrasound (28-33 megahertz, Canon Device) . The cross section area of the nerve will determine . The fascicular organization will be characterized according to 3 types: type 1 (enlarged nerve with hypoechoic nervous fascicles), type 2 (enlarged nerve with the juxtaposition of hypo and hyperechoic fascicles) and type 3 (normal-sized nerve with hypoechoic fascicles poorly differentiated from each other and spiny). Hypervascularity will be evaluated by a doppler signal at the endoneural vessels. The ultrastructural characterization of different types of fascicular organization will also be studied.
Study the relationship between ultrasound data and plasma levels of pro-inflammatory cytokines within the different subgroups of subjects | within 2 months after inclusion
  Serum pro-inflammatory cytokine concentration will be measured using v-plex MSD (Meso Scale Discovery) technology. The ultrasound data taken into account will be the cross section area of the nerve, the echogenicity of the nerve and the presence of hypervascularisation
Study the link between the plasma level of pro-inflammatory cytokines and electrophysiological data obtained by performing electroneurography (ENG) within the different subgroups of subjects | within 2 months after inclusion
  Serum pro-inflammatory cytokine concentration will be measured using v-plex MSD (Meso Scale Discovery) technology. The electrophysiological data will be obtained at the and pre-defined observation sites of the motor nerves: distal latency (in milliseconds); motor conduction velocity (m/s); conduction block: drop in the amplitude and area of the of compound muscle action potential (amplitude in mV).
Study the relationship between ultrasound and electrophysiological data obtained by an electroneurography (ENG) within the different subgroups of subjects | within 2 months after inclusion
  The ultrasound data taken into account will be the cross section area of the nerve, the echogenicity of the nerve and the evaluation of the nerve vascularisation. The electrophysiological data will be obtained at the pre-defined observation site of the motor nerves: distal latency (in milliseconds); motor conduction velocity (m/s);conduction block: drop in the amplitude and area of the compound muscle action potential (amplitude in mV).
Study the relationship between serum concentration of pro-inflammatory cytokines among the different subgroups of patients and clinical scores within different subgroups of subjects using functional assessment scale CMT Neuropathy Score 2 (CMTNS2) | within 2 months after inclusion
  Serum pro-inflammatory cytokine concentration will be measured using v-plex MSD (Meso Scale Discovery) technology.
  The CMT Neuropathy Score 2 (CMTNS2) is a scale used to assess the severity of neuropathy in Charcot-Marie-Tooth disease. The minimum score is 0, indicating no neuropathy, while the maximum score is 36, corresponding to very severe neuropathy. Scores can be divided into four categories: 0 to 4 indicates mild neuropathy, 5 to 14 moderate neuropathy, 15 to 24 severe neuropathy, and 25 to 36 very severe neuropathy. CMTNS2 includes the assessment of sensory symptoms such as paresthesia and pain, motor symptoms such as distal muscle weakness, functional ability based on gait and autonomy, muscle strength, vibration sensitivity, and nerve conduction velocity. This score is used to monitor disease severity
Study the relationship between ultrasound data and the iMAX value: Study the relationship between ultrasound data and IMAX value. | within 2 months after inclusion
  The correlation study between structural changes observed in ultrasound and IMAX values will be conducted as indicated in the previous paragraphs.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Grasse CH, Grasse, Alpes Maritimes
  - Nice CHU, Nice, Alpes Maritimes